CLINICAL TRIAL: NCT00184912
Title: Caffeine Reduces Acute Ischemic Preconditioning
Brief Title: The Effect of Caffeine on Ischemic Preconditioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CAFIRI
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2006-11-29 (Estimated); Status verified 2006-02

CONDITIONS: Caffeine; Ischemic Preconditioning; Ischemia-Reperfusion Injury
MeSH Terms: conditions — Reperfusion Injury | interventions — Caffeine

INTERVENTIONS:
Drug: caffeine
Drug: Technetium-TC99m-labeled Annexin A5
Procedure: ten minutes forearm ischemia
Procedure: ischemic forearm exercise

SUMMARY:
Ischaemic preconditioning (IP) describes the phenomenon that brief periods of ischaemia render the (myocardial) muscle more resistant to a subsequent more prolonged period of ischaemia and reperfusion. Animal studies have provided evidence that adenosine receptor stimulation is an important mediator of IP. As caffeine is an effective adenosine receptor antagonist already at concentrations reached after regular coffee consumption, we aimed to assess whether caffeine impairs IP in humans in vivo. We used a novel and well-validated model to study IP in humans: 99m-Tc-annexin A5 scintigraphy in forearm skeletal muscle.

24 healthy volunteers were randomly assigned to either caffeine (4 mg/kg/iv in 10 minutes) or saline before a protocol for IP.

ELIGIBILITY:
Inclusion Criteria:

* healthy male volunteers

Exclusion Criteria:

-

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24
Dates: Start 2003-09; Study Completion 2006-01

PRIMARY OUTCOMES:
Percentual difference in Annexin A5 targetting between the experimental and control arm one and four hours after intravenous injection.

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Rongen, MD, Phd, Principal Investigator — Radboud University Nijmegen Medical Centre / Department of pharmacology and Toxicology
Locations (1):
- Radboud University Nijmegen Medical Centre / Department of Pharmacology and Toxicology, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Background] Rongen GA, Oyen WJ, Ramakers BP, Riksen NP, Boerman OC, Steinmetz N, Smits P. Annexin A5 scintigraphy of forearm as a novel in vivo model of skeletal muscle preconditioning in humans. Circulation. 2005 Jan 18;111(2):173-8. doi: 10.1161/01.CIR.0000151612.02223.F2. Epub 2004 Dec 27. PMID 15623546
- [Result] Riksen NP, Zhou Z, Oyen WJ, Jaspers R, Ramakers BP, Brouwer RM, Boerman OC, Steinmetz N, Smits P, Rongen GA. Caffeine prevents protection in two human models of ischemic preconditioning. J Am Coll Cardiol. 2006 Aug 15;48(4):700-7. doi: 10.1016/j.jacc.2006.04.083. Epub 2006 Jul 24. PMID 16904537